CLINICAL TRIAL: NCT03152669
Title: The Extended Salford Lung Study ("Ex-SLS") Data Access Project
Status: Recruiting | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 207531
Record Dates: First submitted 2017-05-08; First posted 2017-05-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: asthma; Chronic obstructive pulmonary disease; Salford Lung Study
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic obstructive pulmonary disease: Subjects with COPD who were randomised to treatment in the original SLS
- Asthma: Subjects with asthma who were randomised to treatment in the original SLS.

SUMMARY:
The Salford Lung Study (SLS) subjects represent a group of COPD and asthma patients whose disease is extremely well-characterised over a short time period. Subjects in the SLS originally consented for information relevant to the study to be shared with the sponsor (GSK). These data were limited to three years prior to randomisation and the twelve-month interventional treatment period. Broadened access to patients' data would allow SLS subjects' entire disease journey to be researched, presenting a rare opportunity to improve scientific and clinical understanding of COPD/asthma disease risk, treatment and progression. This proposal seeks to collect additional subject-level data from SLS patients via their electronic medical records (encompassing past and future data for up to 10 years from the date of consent) and via a one-off patient questionnaire administered at the time of consent.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were randomized to treatment in the original SLS studies
* Subjects who are able to, and choose to, provide written consent for the additional information to be collected.

Exclusion Criteria:

* Subjects who were lost to follow-up/moved away, withdrew consent or died during or subsequent to the original SLS studies.
* Subjects considered (at the discretion of the investigator) as too ill to participate or without the mental capacity to provide informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who were randomised for treatment in the original SLS studies
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Retrospective EMR data | Up to 10 years
  All historical data from consent until the beginning of patients' electronic health records, encompassing all routinely-available electronic demographic and health-related data back to a patients' earliest available electronic record.
Prospective EMR data | Up to 10 years
  Prospective longitudinal data, encompassing collection of future routinely-recorded electronic demographic and health-related data for a period of ten years from this consent or until a patient is either lost to follow up or at the time of their death.
Risk factor questionnaire | Up to 10 years
  Historical demographic, COPD/asthma risk factor information and clinical data not routinely available. Collected via paper questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goodall E, Rothnie KJ, Numbere B, Zhang S, Compton C, Wood R, Tritton T, Wild R, Small M, Vestbo J, Woodcock A. Describing the burden of moderate exacerbations in patients with asthma from the Extended Salford Lung Study (Ext-SLS): a retrospective cohort study. Respir Res. 2025 Mar 29;26(1):121. doi: 10.1186/s12931-025-03199-5. PMID 40158113
- [Derived] Meeraus W, Fry M, Yeatman R, Pimenta JM, Astrom J, Barth A, McCorkindale S, Jones R, Leather D. Key Learnings from Running an Extension Study to a Real-World Effectiveness Trial: The Extended Salford Lung Study. Adv Ther. 2021 Sep;38(9):4847-4858. doi: 10.1007/s12325-021-01827-2. Epub 2021 Aug 6. PMID 34357561